CLINICAL TRIAL: NCT06889220
Title: Investigation of Temporomandibular Disorder, Migraine, and Other Related Factors in Patients With Non-Specific Neck Pain
Brief Title: Investigation of Related Factors in Patients With Non-Specific Neck Pain
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Erdi Kayabınar, Assisstant Professor, Hacettepe University
Other Study IDs: 2025/86
Record Dates: First submitted 2025-03-15; First posted 2025-03-21 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Neck Pain
Keywords: non-specific neck pain; temporamandibular joint dysfunction; migraine; Health-related quality of life (HRQoL); Depression
MeSH Terms: conditions — Neck Pain; Migraine Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People with non-specific neck pain: People with non-specific neck pain

SUMMARY:
It has been shown that there is a complex association between neck pain, temporomandibular joint dysfunctions, and migraines, and that these conditions can be influenced by factors such as depression, physical inactivity, and health-related quality of life. Likewise, it is observed that all the factors within this complex structure can actually act as triggers, initiators, or intensifiers of each other.

In recent years, with a more detailed examination of their physiological connections, a reciprocal triangular relationship has been demonstrated between temporomandibular joint (TMJ) dysfunctions, headaches-especially migraines-and neck pain.

A detailed correlation of risk factors affecting neck pain-primarily temporomandibular joint involvement and headaches-in patients with neck pain will help identify underlying secondary effects and facilitate the inclusion of patient-centered, specific exercises in rehabilitation programs for these patients.

Studies in the literature indicate that the relationship between neck pain, temporomandibular joint dysfunctions, and migraines has not been evaluated collectively, and the impact of factors such as depression, physical inactivity, and health-related quality of life on these conditions has not been thoroughly assessed. Therefore, this study aims to comprehensively investigate the effects of temporomandibular joint dysfunctions, migraines, and other associated factors in individuals with non-specific neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18 and 70
* Having non-specific neck pain
* Experiencing migraine-related headaches

Exclusion Criteria:

* Having a diagnosis of cervical trauma, surgery, or disc herniation
* Having a diagnosis of abnormal range of motion in the TMJ or cervical spine, scoliosis, or kyphosis
* Having neurological impairments
* Having systemic diseases
* Having dental or oral pathological lesions, oral infections, facial paralysis, or neuropathic facial pain

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is planned that men and women diagnosed with non-specific neck pain between the ages of 18 and 70 will participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2025-03-19 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index | Baseline
  Neck Disability Index was first defined in 1991. It assesses disability associated with neck pain.
  The index consists of a total of 10 sections, evaluating pain and limitations in activities such as pain, personal care, and lifting, with scores ranging from 0 to 5 for each section. The total score ranges from a minimum of 0 to a maximum of 50. Based on the total score, the classifications are as follows:
  0-4: No disability 5-14: Mild disability 15-24: Moderate disability 25-34: Severe disability 35 and above: Complete disability A validity and reliability study for the Turkish version is available.
Migraine Disability Assessment | Baseline
  The Migraine Disability Assessment Scale (MIDAS) is one of the most commonly used scales for measuring headache-related disability. It assesses migraine-related functional impairment in all activities over the past three months.
  The questionnaire consists of five questions:
  Questions 1, 3, and 5 evaluate the number of days lost due to headaches in the past three months in work or school, household chores, and leisure activities.
  Questions 2 and 4 assess the number of days with reduced productivity at work and in household activities due to headaches.
  The total score is obtained by summing the responses (number of days) for all five questions. The classification based on the total score is as follows:
  0-5 points: Grade I (No or minimal disability) 6-10 points: Grade II (Mild disability) 11-20 points: Grade III (Moderate disability) 21 and above: Grade IV (Severe disability) The Turkish validity and reliability study was conducted.
Helkimo Clinical Dysfunction Index | Baseline
  The ındex was developed in 1974 and evaluates the overall functionality of the craniomandibular region along with TMJ function. It assesses five clinical findings, including:
  1. Mandibular range of motion 2. TMJ function 3. Pain during mandibular movements 4. TMJ pain on palpation 5. Muscle tenderness Each component is scored between 0 and 5.
  1. Assesses limitations in jaw movement, including maximum mouth opening, right and left lateral movements, and forward movement.
  2. component: Evaluates TMJ function by detecting deviations, sounds, and/or joint locking or blockages.
  3. component: Assesses the presence of pain during specific movements.
  4. component: Evaluates muscle pain in the chewing muscles.
  5. component: Assesses discomfort or pain in pre-articular TMJ region through palpation.
  The total score is categorized as follows:
  0 points: No signs or symptoms 1-4 points: Mild dysfunction 5-9 points: Moderate dysfunction 10-25 points: Severe dysfunction

SECONDARY OUTCOMES:
Short Form - 36 | Baseline
  The questionnaire, developed to assess general health status and health-related quality of life, consists of 36 questions and evaluates eight subscales:
  Physical function Physical role Emotional role Energy (vitality) Mental health Social function Pain General health The obtained data are scored between 0 and 100 for each subscale, with higher scores indicating better health status and improved quality of life.
  The Turkish validity and reliability study was conducted.
Beck Depression Inventory | Baseline
  Beck Depression Inventory, developed in 1961, is a 21-item scale assessing depressive symptoms such as pessimism, feelings of failure, lack of satisfaction, guilt, restlessness, fatigue, decreased appetite, indecisiveness, sleep disturbances, and social withdrawal. The validity and reliability study for the Turkish version was conducted in 1988.
  Each item is scored using a four-point Likert scale (0-3), reflecting self-reported experiences of depression-related behaviors. The total score ranges from 0 to 63, with higher scores indicating greater depression severity.
  Score interpretation:
  * Below 10: No or minimal depression
  * 10-18: Mild to moderate depression
  * 19-29: Moderate to severe depression
  * 30-63: Severe depression
International Physical Activity Questionnaire (IPAQ) | Baseline
  The questionnaire consists of seven questions.
  * The first two questions assess vigorous activities
  * The third and fourth questions assess moderate-intensity activities
  * The fifth and sixth questions assess walking
  * The seventh question assesses time spent sitting in the past seven days Based on participants' responses, metabolic equivalent (MET) values are calculated and multiplied by the duration (in minutes and days) to determine the weekly MET-minute score.
  The MET values for different activity levels are:
  * Light activities: 3.3 MET
  * Moderate-intensity activities: 4.0 MET
  * Vigorous activities: 8.0 MET
  Physical activity levels are classified as follows based on total MET-minutes per week:
  * Inactive: less than 600 MET-min per week
  * Low physical activity level: between 600 and 3000 MET-min per week
  * Adequate physical activity level (health-beneficial): more than 3000 MET-min per week.

CONTACTS AND LOCATIONS:
Overall Officials: Erdi KAYABINAR, PhD, Principal Investigator — University of Yalova
Locations (1):
- Yalova university, Yalova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No